CLINICAL TRIAL: NCT06523881
Title: Evaluation of the Effects of Anesthetics and Surgery on Sleep Quality in Patients Undergoing Posterior Spinal Instrumentation Surgery
Brief Title: Effects of Anesthetics and Surgery on Sleep Quality in Patients Undergoing Posterior Spinal Instrumentation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Yücel Bilgin, Orthopedics and Traumatology Surgeon (Spine Surgery), Uludag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UU-YB-2024-01
Record Dates: First submitted 2024-07-12; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Sleep Disturbance; Anesthesia; Adverse Effect
Keywords: posterior instrumentation; sleep quality; anesthetics; spine surgery
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Active Comparator): Group P received propofol Propofol (Propofol-PF® 1% (Polifarma Pharmaceuticals, Tekirdag, Turkey) at a dosage of 75-100 µg/kg/min and remifentanil (Opiva vial®, Tum Ekip Pharmaceuticals Inc., Istanbul, Turkey) IV at a dosage of 0.05-0.2 µg/kg/min.
  Interventions: Procedure: Propofol (Propofol-PF® 1% (Polifarma Pharmaceuticals, Tekirdag, Turkey)
- Group S (Active Comparator): Group S utilized sevoflurane (Sevorane® liquid 100%, Abbvie Pharmaceuticals, Istanbul, Turkey) for anesthesia maintenance, with an end-tidal sevoflurane concentration ranging from 1 to 1.5 minimal alveolar concentrations. Furthermore, remifentanil (Opiva vial®, Tum Ekip Pharmaceuticals Inc., Istanbul, Turkey) was administered IV at an infusion rate ranging from 0.05 to 0.2 µg kg/min.
  Interventions: Procedure: Sevoflurane (Sevorane® liquid 100%, Abbvie Pharmaceuticals, Istanbul, Turkey)

INTERVENTIONS:
Procedure: Sevoflurane (Sevorane® liquid 100%, Abbvie Pharmaceuticals, Istanbul, Turkey) — Sevoflurane (Sevorane® liquid 100%, Abbvie Pharmaceuticals, Istanbul, Turkey) is a medication used during anesthesia. It is administered by inhalation with an anesthesia device.
  Arms: Group S
Procedure: Propofol (Propofol-PF® 1% (Polifarma Pharmaceuticals, Tekirdag, Turkey) — Propofol is a drug used during anesthesia. It is administered intravenously using an infusion pump during surgical procedures.
  Arms: Group P

SUMMARY:
Investigators aimed to evaluate the impact of the anesthesia method and surgical procedure on the sleep patterns and sleep quality of patients undergoing posterior spinal instrumentation using the Pittsburgh Insomnia Rating Scale-20 (PIRS-20).

DETAILED DESCRIPTION:
A total of 40 participants ASA (American Society of Anesthesiology) I-III aged 18 and over who underwent elective spinal posterior instrumentation was included. The participants were divided into two groups randomly - those with sevoflurane and remifentanil anesthesia and those with total intravenous anesthesia (TIVA) - using the closed envelope method. Participants were evaluated before and after the surgery with the PIRS-20 (surgery one month previously and postoperative 7th day) for sleep quality, VAS (Visual Analogue Scale; recorded preoperative night and postoperative first hour), pain, and State-Trait Anxiety Inventory (STAI) for anxiety (recorded preoperative night and postoperative 7th day) scores.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiology) I-III
* Aged 18 and over
* Who underwent elective spinal posterior instrumentation

Exclusion Criteria:

* Aged 17 and under
* ASA (American Society of Anesthesiology) IV
* Presence of psychological illness
* Presence of psychological illness
* Presence of sleep disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Insomnia Rating Scale-20 | Preoperative one month
  Sleep score: Minimum value:0 Maximum value:60 Higher scores mean a worse outcome.
Pittsburgh Insomnia Rating Scale-20 | Postoperative seventh day
  Sleep score: Minimum value:0 Maximum value:60 Higher scores mean a worse outcome.
Visual Analogue Scale | Preoperative one day
  Pain score: Minimum value:0 Maximum value:10 Higher scores mean a worse outcome.
Visual Analogue Scale | Postoperative first hour
  Pain score: Minimum value:0 Maximum value:10 Higher scores mean a worse outcome.
State-Trait Anxiety Inventory | Preoperative one day
  Anxiety score: Minimum value:20 Maximum value:80 Higher scores mean a worse outcome.
State-Trait Anxiety Inventory | Postoperative seventh day
  Anxiety score: Minimum value:20 Maximum value:80 Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yücel Bilgin, MD, Principal Investigator — Uludag University
Locations (1):
- Uludag University, Bursa, Nilufer, Turkey (Türkiye)